CLINICAL TRIAL: NCT06123507
Title: A Randomized Pragmatic Feasibility Trial to Promote Student Perspective-Taking on Client Physical Activity: A Collaborative Project
Brief Title: A Pragmatic Feasibility Trial to Promote Student Perspective-Taking on Client Physical Activity: A Collaborative Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E2018:008; 48798 (Other Grant/Funding Number: University of Manitoba); 322464 (Other Grant/Funding Number: Manitoba Centre for Nursing and Health Research)
Record Dates: First submitted 2023-10-11; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Communication
Keywords: Perspective-taking; Empathy; Education; Feasibility
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: This randomized mixed-methods parallel two-arm feasibility trial used a 1:1 allocation ratio in Excel. This study's primary purpose was to assess the feasibility, appropriateness, and acceptability of a randomized pilot trial where some health-care students received a Full educational Intervention on perspective-taking and others received a Partial Intervention.
Who Masked: Outcomes Assessor
Masking Description: Client-actors were masked to condition. Investigators were masked while determining participants' perceptual understanding scores (i.e., how accurate participants were at inferring the client-actor's thoughts and feelings). In-lab research assistants were not masked to condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full educational intervention condition (Experimental): The Full intervention condition included a perspective-taking workshop plus independent practice and video-feedback
  Interventions: Behavioral: Student practitioner perspective-taking intervention
- Partial intervention condition (Active Comparator): The Partial intervention condition involved video-feedback alone. In this condition, participants were provided with a link to the perspective-taking workshop after the study was complete.
  Interventions: Behavioral: Student practitioner perspective-taking intervention

INTERVENTIONS:
Behavioral: Student practitioner perspective-taking intervention — This intervention compares the outcomes where some learn about and practice perspective-taking and others do not. All participants received at least a partial intervention through getting video-feedback on their dialogue with a client actor.

SUMMARY:
This mixed-methods parallel two-arm trial assessed the feasibility, appropriateness, and acceptability of a theoretically-informed intervention designed to improve perspective-taking skills in preparation for a future definitive randomized control trial. Using a 1:1 allocation ratio, student participants (N = 163) in Respiratory, Physical, and Occupational Therapy; Nurse Practitioner; and Kinesiology programs at a Canadian university were randomly assigned to full or partial intervention conditions. Full intervention participants completed an online workshop on perspective-taking and practiced perspective-taking prior to an in-lab 10-minute dialogue with a trained client-actor (masked to condition) about the actor's physical inactivity. Partial intervention participants received the workshop after the dialogue, and were instructed to be aware and mindful of the approach that they took to seek understanding. To be considered feasible, outcomes needed to meet or surpass our criteria (e.g., within-course recruitment: 85-95% of a course when embedded within a course, 5-10% when not embedded). Feasibility and appropriateness were assessed by comparing recruitment rates, protocol, and psychometric outcomes to criteria. Acceptability was assessed by analyzing exit interviews. Recruitment rates, protocol, and psychometric outcomes largely met criteria, and the study was acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Must be a student at the University of Manitoba
* Must have completed course content on behaviour change communication

Exclusion Criteria:

* Full intervention participants were excluded from descriptive statistics calculations if they partially completed the workshop or did not complete all phases due to client-actor availability
* Data from participating in additional study sessions were excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Recruitment rate when embedded within a course | Within 2 years of study commencement (February 2018 - December 2019)
  85-95% recruitment rate
Recruitment rate when not embedded within a course | Within 2 years of study commencement (February 2018 - December 2019)
  5-10% recruitment rate
Recruitment time | Within 2 years of study commencement (February 2018 - December 2019)
  Time to finish recruiting in years
Program recruitment | Within 2 years of study commencement (February 2018 - December 2019)
  Count of number of participants per program
Workshop completion | Prior to in-lab participation
  Percent that completed all pages of the workshop
Practice time length | Prior to in-lab participation
  Time in weeks
Adherence for not making a plan of action with the client-actor | Through in-lab completion, an expected average of 2 hours
  Percent that adhered to instructions
Lab session length | Through in-lab completion, an expected average of 2 hours
  Average lab session length, and time participants spent in the lab in hours and minutes
Employee training | Through study completion, up to 2 years
  Time in hours
Appropriateness of measure means as assessed by examining data for floor and ceiling effects | Post study completion, after 2 years
  A scale mean will be created for all measures. To assess appropriateness for inclusion in the definitive trial, we will examine the means for floor and ceiling effects. There should be no evidence of floor or ceiling effects in study measures. If there is evidence of extreme means, then we will consider a different measure for the definitive trial.
Amount of missing data | Post study completion, after 2 years
  To assess appropriateness for inclusion in the definitive trial, the amount of missing data will be examined for each measure. There should be no more than 5% for each study measure. If there is evidence of excessive missing data for a measure, then we will consider a different measure for the definitive trial.
Appropriateness of Cronbach's alpha as assessed by an alpha above .70 for each measure | Post study completion, after 2 years
  To assess appropriateness for inclusion in the definitive trial, we will calculate Cronbach's alpha for each measure. Cronbach's alpha should be at least .70 for each study measure. If there is evidence of low Cronbach's alpha for a measure, then we will consider a different measure for the definitive trial.

SECONDARY OUTCOMES:
Instructor interest | At time of contact through study completion, up to 2 years
  Count of instructors who express interest in the study
Integration rate | Prior to the study period
  Count of how many instructors embedded the course into their study
Participant demographics | At baseline
  Counts and percentages
Prior communication training | At baseline
  Counts and percentages for self-reported training
Acceptability | Post study completion, after 2 years
  Examining exit interviews and field notes using manifest content analysis and constant comparison techniques

CONTACTS AND LOCATIONS:
Overall Officials: Shaelyn Strachan, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
The data will not be shared. The data are not publicly available because we did not get permission from participants.

REFERENCES:
- [Derived] Hoplock LB, Lobchuk MM, Strachan SM, Halas G, Olfert C, Webber S, Parsons JL. A randomized pragmatic feasibility trial to promote student perspective-taking on client physical activity level: a collaborative project. Pilot Feasibility Stud. 2024 Sep 28;10(1):123. doi: 10.1186/s40814-024-01547-8. PMID 39342378